CLINICAL TRIAL: NCT04560166
Title: Naxitamab and Granulocyte-Macrophage Colony Stimulating Factor in Combination With Irinotecan and Temozolomide in Patients With High-Risk Neuroblastoma With Primary Refractory Disease or in First Relapse. An International, Single-Arm, Multicenter Phase 2 Trial.
Brief Title: Naxitamab and GM-CSF in Combination With IT in Patients With High-Risk Neuroblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to business priorities
Sponsor: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 203
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-02

CONDITIONS: Neuroblastoma Recurrent
MeSH Terms: interventions — naxitamab; Granulocyte-Macrophage Colony-Stimulating Factor; Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Naxitamab and GM-CSF in combination with irinotecan and temozolomide (Experimental): A treatment cycle is 21 days. The patients will receive irinotecan 50 mg/m2/day IV and temozolomide 100 mg/m2/day orally (both on Days 1-5) in combination with naxitamab 2.25 mg/kg/day IV (Days 2, 4, 8 and 10) (total 9 mg/kg per cycle), and GM-CSF 250 ug/m2/day sc, (Days 6-10).
  Patients will receive up to 18 IT cycles after enrollment. Naxitamab and GM-CSF will be given for at least 8 cycles.
  Interventions: Drug: Naxitamab and GM-CSF in combination with irinotecan and temozolomide

INTERVENTIONS:
Drug: Naxitamab and GM-CSF in combination with irinotecan and temozolomide — * Irinotecan, solution for infusion (20 mg/mL)
  * Temozolomide, capsules (5 mg, 20 mg and 100 mg)
  * The humanized immunoglobulin isotype G (IgG1) monoclonal antibody (mAb) naxitamab, solution for infusion (4 mg/mL)
  * Sargramostim (GM-CSF), lyophilized 250 µg single use vial (250 µg/vial)

SUMMARY:
An International, Single-Arm, Multicenter Phase 2 Trial.

DETAILED DESCRIPTION:
This is an international, single-arm, multicenter phase 2 trial, in patients ≥ 12 months of age with high-risk NB with primary refractory disease or in first relapse. Patients will receive naxitamab + GM-CSF + irinotecan/temozolomide. The Follow-Up period ends 2 years after End of Treatment.

ELIGIBILITY:
Inclusion Criteria:

* Neuroblastoma (NB)
* Documented high-risk disease
* Receipt of Standard of Care (SoC) frontline induction/consolidation therapy (including surgery, chemotherapy, ASCT, MIBG, radiotherapy, immunotherapy, or retinoids)
* Active disease despite previous aggressive multi-drug chemotherapy, defined as one of the following:

  * verified first progression during multi-drug frontline treatment or
  * verified first episode of relapse, defined as recurrence after response to frontline treatment, or
  * verified first designation of refractory disease, defined as persistent metastatic disease (SD or minor response by INRC and MIBG curie score ≥3) detected at conclusion of at least 4 cycles of multi-drug induction chemotherapy on or according to a high-risk NB treatment protocol as defined above
* The patients must have one of the following (locally assessed) obtained within 3 weeks prior to enrollment and at least 10 calendar days after end of any prior anti-cancer treatment:

  * Measurable tumor on CT/MRI scan that is MIBG-avid or demonstrates increased FDG uptake on PET scan
  * MIBG (Metaiodobenzylguanidine) scan with positive uptake at a minimum of one site. This site must represent disease recurrence after completion of therapy, progressive disease on therapy, or refractory disease during induction
* Age ≥ 12 months at enrollment
* Written informed consent

Exclusion Criteria:

* Myelodysplastic syndrome or any malignancy other than NB
* Any systemic anti-cancer therapy within 3 weeks
* Autologous stem cell transplant (ASCT) within 6 weeks prior to enrollment or ongoing toxicity due to the stem cell transplant at the discretion of the investigator
* Therapeutic 131I-MIBG within 6 weeks prior to enrollment
* Radiotherapy (RT) within 4 weeks prior to enrollment at any lesion site that will be identified as a target lesion to measure tumor response
* Prior treatment with anti-GD2 if the patient experienced Progressive Disease (PD) while on anti-GD2 treatment
* Receipt of second line chemotherapy after designation of primary refractory disease or first relapse or PD
* NB in Bone Marrow (BM) only
* NB in the Central Nervous System (CNS) or leptomeningeal disease within 6 months prior to enrollment
* Performance status of < 50% as per the Lansky scale (patients less than 16 years of age) or Karnofsky scale (for patients aged 16 years or older)
* Life expectancy of less than 6 months
* Left ventricular ejection fraction < 50% by echocardiography
* Inadequate pulmonary function
* Diarrhea Grade ≥ 2
* Treatment with long-acting myeloid growth factor within 14 days or short-acting myeloid growth factor within 7 days prior to first dose of GM-CSF
* Receipt of immunosuppressive treatment (local steroids excluded) within 4 weeks prior to enrollment
* Life threatening infection(s)
* Uncontrolled seizure disorders despite anticonvulsant therapy (defined as a seizure event within 3 months prior to enrollment)
* Treatment with enzyme-inducing anticonvulsants including phenytoin, phenobarbital, or carbamazepine for at least 7 days prior to enrollment
* Concomitant use with St John's wort
* Allogeneic hematopoietic stem cell transplantation (allo-SCT) or donor-lymphocyte-infusion (defined as any kind of active allogeneic lymphocyte suspension)
* Treatment with Hematopoietic Progenitor Cell (HPC) boost within 2 months prior to enrollment
* History of allergy or known hypersensitivity to GM-CSF, yeast-derived products, or any component of GM-CSF, naxitamab, irinotecan or temozolomide
* History of anaphylactic reactions CTCAE Grade 4 related to prior anti-GD2 antibody therapy
* Unacceptable hematological status at screening, defined as one of the following:

  * Hemoglobin <5.0 mmol/L (<8 g/dL)
  * White blood cell count <1000/µL
  * Absolute neutrophil count <750/µL
  * Platelet count < 75,000/µL
* Unacceptable liver function at screening, defined as one of the following:

  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >5 times upper normal limit (UNL)
  * Total bilirubin >1.5 x UNL
* Unacceptable kidney function at screening, defined as estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 calculated by the 2009 revised Bedside Schwartz Equation
* Inability to comply with protocol
* Significant intercurrent illness (any ongoing serious medical problem unrelated to cancer or its treatment) that is not covered by the detailed exclusion criteria and that is expected to interfere with the action of trial agents or to significantly increase the severity of the toxicities experienced from trial treatment
* Females of childbearing potential who are pregnant, breast feeding, intend to become pregnant, or are not using adequate contraceptive methods or males who are not using adequate contraceptive methods

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Hong Kong Children's Hospital, Hong Kong, Hong Kong
- South Korea (2):
  - Asan Medical Center Children's Hospital, Seoul
  - Seoul National University Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- Naxitamab and GM-CSF in Combination With Irinotecan and Temozolomide: A treatment cycle is 21 days. The patients will receive irinotecan 50 mg/m2/day IV and temozolomide 100 mg/m2/day orally (both on Days 1-5) in combination with naxitamab 2.25 mg/kg/day IV (Days 2, 4, 8 and 10) (total 9 mg/kg per cycle), and GM-CSF 250 ug/m2/day sc, (Days 6-10).
  Patients will receive up to 18 IT cycles after enrollment. Naxitamab and GM-CSF will be given for at least 8 cycles.
  Naxitamab and GM-CSF in combination with irinotecan and temozolomide: • Irinotecan, solution for infusion (20 mg/mL)
  * Temozolomide, capsules (5 mg, 20 mg and 100 mg)
  * The humanized immunoglobulin isotype G (IgG1) monoclonal antibody (mAb) naxitamab, solution for infusion (4 mg/mL)
  * Sargramostim (GM-CSF), lyophilized 250 µg single use vial (250 µg/vial)
Period: Overall Study
Arm/Group | Naxitamab and GM-CSF in Combination With Irinotecan and Temozolomide
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Naxitamab and GM-CSF in Combination With Irinotecan and Temozolomide
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 4.5 [4 to 5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: The proportion of patients obtaining a centrally assessed complete response (CR) or partial response (PR) according to the International Neuroblastoma Response Criteria (INRC)
Time Frame: 84 days
Population: The trial was terminated prematurely and no results from primary or secondary efficacy outcomes are available because images and bone marrow pathology were never submitted for central response assessment.
Arm/Group | Naxitamab and GM-CSF in Combination With Irinotecan and Temozolomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From day of first IMP administration until 42 days after last IMP administration, an average of 34 weeks.
Arm/Group | Naxitamab and GM-CSF in Combination With Irinotecan and Temozolomide
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naxitamab and GM-CSF in Combination With Irinotecan and Temozolomide (N=2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naxitamab and GM-CSF in Combination With Irinotecan and Temozolomide (N=2)
Anaemia (Blood and lymphatic system disorders) | 2 (8)
Abdominal pain (Gastrointestinal disorders) | 1 (30)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (4)
Fatigue (General disorders) | 1 (1)
Localised oedema (General disorders) | 1 (1)
Pain (General disorders) | 1 (27)
Pyrexia (General disorders) | 2 (7)
Swelling (General disorders) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (18)
Platelet count decreased (Investigations) | 1 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (24)
Hypotension (Vascular disorders) | 2 (19)

LIMITATIONS AND CAVEATS:
Terminated due to business priorities resulting from slow recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT04560166/Prot_SAP_000.pdf